CLINICAL TRIAL: NCT05894031
Title: The Effectiveness of the Wim Hof Method on Cardiac Autonomic Function, Blood Pressure, Arterial Compliance, and Different Psychological Parameters
Brief Title: The Effectiveness of the Wim Hof Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-04-00004
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Healthy; Blood Pressure; Cold Exposure; Stress
Keywords: Blood pressure; Hemodynamics; Heart rate variability; Perceived stress; Meditation; Cold exposure; Breathing-method

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with parallel arms
Who Masked: Outcomes Assessor
Masking Description: Blinding of outcome assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group was instructed to perform the Wim Hof Method daily over the course of 15 days. The participants could choose when to do so throughout the day, however, the components were to be performed in a strict, sequential order: breathing exercises, followed by meditation, and then cold exposure. Participants were asked to complete a daily log in which they documented whether they performed the procedure and for how long. Altogether, the procedure lasted about 15 minutes.
  Interventions: Behavioral: Wim Hof Method
- Control (No Intervention): The control group received noch intervention throughout the intervention period.

INTERVENTIONS:
Behavioral: Wim Hof Method — The intervention followed the guidelines provided by Wim Hof. The intervention comprised three components: cold water exposure, breathing exercise, and meditation.The participants were instructed to perform the WHM daily over the course of 15 days. The participants could choose when to do so throughout the day, however, the components were to be performed in a strict, sequential order: breathing exercises, followed by meditation, and then cold exposure. Participants were asked to complete a daily log in which they documented whether they performed the procedure and for how long. Altogether, the procedure lasted about 15 minutes.
  Arms: Intervention

SUMMARY:
The Wim Hof Method is a multi-disciplinary approach to physical and mental well-being combining cold exposure, breathing exercises, and meditation. This study evaluated the effects of a 15-day WHM intervention on cardiovascular parameters at rest and during a cold pressor test, as well as on various psychological parameters.

DETAILED DESCRIPTION:
The Wim Hof Method (WHM) is a multi-disciplinary approach to physical and mental well-being combining cold exposure, breathing exercises, and meditation. This study evaluated the effects of a 15-day WHM intervention on cardiovascular parameters at rest and during a cold pressor test (CPT), as well as on various psychological parameters.

42 participants were randomized into an intervention (IG) and a control (CG) group. Throughout the 15-day intervention, the IG performed the WHM daily. The intervention followed the guidelines provided by Wim Hof. The intervention comprised three components: cold water exposure, breathing exercise, and meditation. The participants were instructed to perform the WHM daily over the course of 15 days. The participants could choose when to do so throughout the day, however, the components were to be performed in a strict, sequential order: breathing exercises, followed by meditation, and then cold exposure. Participants were asked to complete a daily log in which they documented whether they performed the procedure and for how long. Altogether, the procedure lasted about 15 minutes. The CG did not receive an intervention throughout the intervention period.

Before and after the intervention, systolic (SBP) and diastolic blood pressure (DBP), pulse wave velocity (PWV), heart rate (HR), root mean sum of squared distance (RMSSD), and standard deviation of intervals between successive heartbeats (SDNN) were assessed at rest and during a CPT. Furthermore, perceived stress (PSS), positive affect (PANAS+), negative affect (PANAS-), and subjective vitality (trait (SVSt) and state (SVSs)) was determined.

ELIGIBILITY:
Inclusion Criteria:

* Being male
* No underlying health conditions
* Not using antihypertensive or other cardiovascular medications
* Not engaging in regular exercise training
* Written informed consent

Exclusion Criteria:

* Having prior experience with any of the components of the intervention (breathing, meditation, or cold exposure)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male participants were eligible for the study.
Enrollment: 42 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean systolic blood pressure | 15 days
  Participants were instructed to rest in a supine position for 10 minutes prior to the measurement. At least two readings were taken on the right upper arm, using custom-fitted arm cuffs.
Change from baseline in the mean diastolic blood pressure | 15 days
  Participants were instructed to rest in a supine position for 10 minutes prior to the measurement. At least two readings were taken on the right upper arm, using custom-fitted arm cuffs.

SECONDARY OUTCOMES:
Change from baseline in the mean pulse wave velocity | 15 days
  Participants were instructed to rest in a supine position for 10 minutes prior to the measurement. At least two readings were taken on the right upper arm, using custom-fitted arm cuffs.
Change from baseline in the mean heart rate variability | 15 days
  Heart rate variability (HRV) was measured using a heart rate monitor and chest strap. Participants were instructed to empty their bladder before the measurement, which was conducted after a 5-minute supine rest period with a stabilized HRV signal. The measurement consisted of a 5-minute recording of intervals between successive heartbeats at a 1000 Hz sampling rate. Participants were instructed to breathe normally, remain quiet, and maintain a calm state throughout the measurement.
Change from baseline in positive affect | 15 days
  The German version of the Positive and Negative Affect Schedule was used.
Change from baseline in negative affect | 15 days
  The German version of the Positive and Negative Affect Schedule was used.
Change in subjective vitality | 15 days
  The German 6-item Version of the Subjective Vitality Scale was used.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Ketelhut, PhD, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All raw data are available on request to the corresponding author.
Supporting Information: Study Protocol, ICF
Time Frame: After the publication of the results for 5 years.
Access Criteria: PErsonal contact with corresponding author.

REFERENCES:
- [Derived] Ketelhut S, Benzing V, Zehnder C, Amor L, Schurch Y, Burger M, Schmid S, Nigg CR. Effects of exergaming versus endurance training on cardiorespiratory fitness and hemodynamic parameters: a randomized controlled trial. Eur J Appl Physiol. 2025 Jul;125(7):1817-1830. doi: 10.1007/s00421-025-05743-z. Epub 2025 Mar 11. PMID 40067458